CLINICAL TRIAL: NCT06210620
Title: Prospective, Observational Registry to Collect Standard of Care Clinical Testing Data From Lower-limb Prosthesis Patients Via the PRO App.
Brief Title: Pro APP Prosthetic Outcome Registry
Status: Recruiting | Type: Observational
Sponsor: Össur Iceland ehf (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP2023092221
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-03

CONDITIONS: Amputation
Keywords: Registry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
A national, multi-center registry of patients using lower-limb prosthesis, their profiles and devices, and their long-term follow-up and clinical outcomes.

DETAILED DESCRIPTION:
This US national patient and outcome registry will provide demographic information on lower-limb prosthesis users and their real-world clinical outcomes. The intent is to collect data from multiple certified O&P clinics that have access to use the digital data collection tool PRO App (https://www.ossur.com/en-us/professionals/PRO App). Any patient undergoing prosthetic treatment with their prescribed devices (such as a new fitting, alignment, or replacement of a previous prosthesis) at the investigational sites will be offered to provide data to the registry. Data collection will be a part of the standard of care and is entered by the participating prosthetists, physicians, physical therapists, or other designated staff during clinic/service visits. Data already entered into the PRO App system may also be collected into the registry if the participant consents. This registry will recruit patients who meet the inclusion criteria. Participation is fully voluntary. After the enrollment, all participants would be evaluated during follow-up visits as demanded by their standard of care.

Exploratory analyses may be implemented, utilizing the already collected data, to investigate specific populations and their outcomes depending on the enrollment of said population groups. As an example; data will be collected from the registry to stratify two demographically matching groups of prosthetic users using a powered knee and a non-powered knee.

ELIGIBILITY:
Inclusion Criteria:

Cognitive ability to understand all instructions and questionnaires in the study Willing and able to participate in the study and follow the protocol Individuals with lower limb loss, amputation or deficiency

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient undergoing lower limb prosthetic treatment with their prescribed devices, such as a new fitting, alignment, or replacement of a previous prosthesis.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2033-09 (Estimated); Study Completion 2033-09 (Estimated)

PRIMARY OUTCOMES:
Provide data on patient characteristics | 10 years
  The primary objective of this study is to generate a national, multi-center registry of patients using lower-limb prosthesis, their profiles and devices, and their long-term follow-up and clinical outcomes.

SECONDARY OUTCOMES:
Provide data on device performance | 10 years
  To perform comparative analysis on the population and subgroups based on demographics, device brands, device types, device technology, patient reported outcomes, observer-reporter, and objective clinical assessments

CONTACTS AND LOCATIONS:
Locations (1):
- Össur Americas, Irvine, California, United States